CLINICAL TRIAL: NCT02953925
Title: National-wide Survey on Primary Health Care in China
Acronym: China-PHC
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHC Survey
Record Dates: First submitted 2016-10-30; First posted 2016-11-03 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Primary Health Care
Keywords: primary health care; village doctor; township hospital; community health center

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- primary health care users: Subjects with high risk of cardiovascular diseases who lived in the catchment areas of the participating PHC institutions.

SUMMARY:
The survey aims to support health policy making, this survey aims to comprehensively assess the capability and quality of PHC in different regions in China. The study is based on the China PEACE MPP network, including about 4000 rural and urban primary health care institutions scattered over 31 provinces in Mainland China. The investigators intended to enroll about 30,000 PHC healthcare providers. Meanwhile, the investigators drew a random samples (>50,000) of patients from MPP high-risk of CVD population. In this survey, data on structure, process, and outcome of PHC system in China will be collected by questionnaires, specified by organization, healthcare providers and patients. Meanwhile, the investigators will collect the original documents from participating PHC institutions, covering the aspects of finance, employment, essential medical list (EMS), public health service report and prescriptions. The investigators will analyze data in align with key indicators, to assess the capability and quality of PHC across different regions in China.

DETAILED DESCRIPTION:
The survey aims to support health policy making, this survey aims to comprehensively assess the capability and quality of PHC in different regions in China. The study is based on the China PEACE MPP network, including about 4000 rural and urban primary health care institutions scattered over 31 provinces in Mainland China. The investigators intended to enroll about 30,000 PHC healthcare providers. Meanwhile, the investigators drew a random samples (>50,000) of patients from MPP high-risk of CVD population. In this survey, data on structure, process, and outcome of PHC system in China will be collected by questionnaires, specified by organization, healthcare providers and patients. Meanwhile, the investigators will collect the original documents from participating PHC institutions, covering the aspects of finance, employment, essential medical list (EMS), public health service report and prescriptions. The investigators will analyze data in align with key indicators, to assess the capability and quality of PHC across different regions in China.

1. PHC organizations: All rural and urban PHC institutions in the MPP network are invited to participate the survey. The MPP identified the eligible collaborating institutions based on the amount of residents in the catchment area, population stability, economic condition and geographic location.
2. PHC providers: The investigators intended to invite all the healthcare providers who work in the participating PHC institutions to participate the survey. In this survey, healthcare workers refer to physicians, nurses, public health workers and village doctors based on their professional education background. The village doctors are those who work in the village clinics with a certificate of village doctor.
3. Patients: The investigators intended to interview patients, who lived in the catchment areas of the participating PHC institutions, to study the satisfaction on the PHC services and health insurance, health outcomes and out-of-pocket payment for the services.

ELIGIBILITY:
Inclusion Criteria:

* lived in the catchment areas of the participating PHC institutions
* aged 35-75 years
* screened in China PEACE MPP project
* with high risk for cardiovascular diseases

Exclusion Criteria:

-

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects identified as high risk for cardiovascular diseases in China PEACE MPP study, who lived in the catchment areas of the participating PHC institutions
Sampling Method: Probability Sample
Enrollment: 50000 (Actual)
Dates: Start 2016-11; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Use of on the PHC services | 1 year
  Subjects' experiences of seeking PHC is collected using a self-administrative questionnaire. Also, the investigators will extract information from original documents from PHC institusions, covering the aspects of finance, employment, essential medical list (EMS), public health service report and prescriptions

SECONDARY OUTCOMES:
Satisfaction on the PHC services | 1 year
  Subjects' opinion on PHC is collected using a self-administrative questionnaire

IPD SHARING:
Plan to Share IPD: Undecided